CLINICAL TRIAL: NCT00252707
Title: A Multicentre, Randomised, Open-Label, Parallel-Group, Phase III Post-Marketing Clinical Study to Compare the Overall Survival Between Gefitinib and Docetaxel in Patients With Advanced or Metastatic (Stage IIIB/IV), or Recurrent Non-Small Cell Lung Cancer, Who Have Failed One or Two Chemotherapy Regimens
Brief Title: Iressa 2nd Line Phase III Study in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D791AL00001; V-15-32
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Docetaxel

INTERVENTIONS:
Drug: Gefitinib or Docetaxel

SUMMARY:
In this study, among the patients with non-small cell lung cancer, those with metastasis or recurrence and previous treatment with chemotherapy will receive gefitinib or docetaxel, and we will compare the effectiveness and safety of gefitinib with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* You are "histologically" or "cytologically" confirmed to have recurrent or metastatic NSCLC
* You have been treated with chemotherapy including platinums for NSCLC.

Exclusion Criteria:

* You have received treatment for non-small lung cancer within 4 weeks before your participation in this study (except for specific therapies)
* You have or had any disease of acute lung injury, idiopathic pulmonary fibrosis, pulmonary pneumonia, or pneumoconiosis evident on the X-ray
* You have or had any disease of radiation pneumonia or drug-induced pneumonia, which requires treatment with corticosteroids

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2003-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Determine the overall survival with these treatments as the primary outcome.

SECONDARY OUTCOMES:
Determine the followings as the secondary outcome variables:
- Progression-free survival (PFS)
- Time to treatment failure (TTF)
- Objective tumour response (CR, PR) and the disease control rate (CR, PR, SD [≥12 weeks]) based on the RECIST guidelines
- Lung cancer subscale (LCS)
- QOL according to FACT-L questionnaire
- Frequency and severity of adverse events.
Determine the followings as the exploratory outcome variables:
- Biomarkers related to expression, activation and dimerisation of EGFR and other ErbB family receptors and associated pathways including downstream signalling pathways
- Biomarkers related to somatic (non-inheritable) mutation analyses of genes of the ErbB family, their signalling pathways and associated pathways which are thought to be influenced by gefitinib in tumour cells.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director, MD, Study Director — AstraZeneca
Locations (40):
- Japan (40):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Okazaki, Aichi-ken
  - Research Site, Hirosaki, Aomori
  - Research Site, Kashiwa, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Gifu, Gifu
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Akashi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Naka-gun, Ibaraki
  - Research Site, Isehara, Kanagawa
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Sendai, Miyagi
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Ōmura, Nagasaki
  - Research Site, Niigata, Niigata
  - Research Site, Beppu, Oita Prefecture
  - Research Site, Okayama, Okayama-ken
  - Research Site, Habikino, Osaka
  - Research Site, Izumisano, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Sayama, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Iwata, Shizuoka
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Chūō, Tokyo
  - Research Site, Kiyose, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Sumida City, Tokyo
  - Research Site, Toshima-ku, Tokyo
  - Research Site, Yamagata, Yamagata
  - Research Site, Ube, Yamaguchi
  - Research Site, Kanazawa

REFERENCES:
- [Derived] Maruyama R, Nishiwaki Y, Tamura T, Yamamoto N, Tsuboi M, Nakagawa K, Shinkai T, Negoro S, Imamura F, Eguchi K, Takeda K, Inoue A, Tomii K, Harada M, Masuda N, Jiang H, Itoh Y, Ichinose Y, Saijo N, Fukuoka M. Phase III study, V-15-32, of gefitinib versus docetaxel in previously treated Japanese patients with non-small-cell lung cancer. J Clin Oncol. 2008 Sep 10;26(26):4244-52. doi: 10.1200/JCO.2007.15.0185. PMID 18779611